CLINICAL TRIAL: NCT03720522
Title: The Bern Heart and Brain Interaction Study - Interaction Between Brain and Heart in Acute Ischemic Stroke
Acronym: BEHABIS
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01087
Record Dates: First submitted 2018-10-11; First posted 2018-10-25 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Patients suffering from acute myocardial infarction: Patients with positive gadolinium late enhancement and positive intramyocardial oedema in the short CMR have an acute myocardial infarction and will be allocated to group 1.
  Interventions: Procedure: Short cardiovascular MRI (CMR); Procedure: Blood draw; Procedure: Urine (collection over 24h)
- Group 2: Patients suffering from chronic myocardial infarction: Patients with elevated (≥ 0.015 mg/L) high sensitive troponin T (hsTnT) levels, positive gadolinium late enhancement and/or positive myocardial infarction suffer from chronic myocardial infarction or significant coronary stenosis. They will be allocated to group 2 and receive coronary angiography in a timely manner according to clinical routine and current guidelines.
  Interventions: Procedure: Short cardiovascular MRI (CMR); Procedure: Adenosine-perfusion cardiovascular MRI (CMR); Procedure: Blood draw; Procedure: Urine (collection over 24h)
- Group 3: Patients suffering from stunned neurogenic myocardium: Patients with elevated (≥ 0.015 mg/L) high sensitive troponin T (hsTnT) levels and presence of wall motion abnormalities (WMA) have potential WMA due to neurogenic myocardial stunning. They will be allocated to group 3.
  These patients will undergo a follow-up CMR without adenosine-perfusion after 3 months to confirm improvement/normalization of WMA.
  Patients with normal (< 0.015mg/L) hsTnT levels and presence of WMA will also be allocated to group 3.
  Interventions: Procedure: Short cardiovascular MRI (CMR); Procedure: Adenosine-perfusion cardiovascular MRI (CMR); Procedure: Blood draw; Procedure: Urine (collection over 24h)
- Group 4: Control: Patients with normal (< 0.015mg/L) high sensitive troponin T (hsTnT) levels without late enhancement, without myocardial infarction and without wall motion abnormalities will serve as control group and will be classified to group 4.
  Interventions: Procedure: Short cardiovascular MRI (CMR); Procedure: Adenosine-perfusion cardiovascular MRI (CMR); Procedure: Blood draw; Procedure: Urine (collection over 24h)

INTERVENTIONS:
Procedure: Short cardiovascular MRI (CMR) — A short CMR without additional contrast administration will be performed immediately after the routine brain MRI (at admission or after 24h).
Procedure: Adenosine-perfusion cardiovascular MRI (CMR) — An adenosine-perfusion CMR using contrast medium (gadolinium) will be performed in all patients (except group 1) between 48h and 6 days after admission.
  Groups: Group 2: Patients suffering from chronic myocardial infarction; Group 3: Patients suffering from stunned neurogenic myocardium; Group 4: Control
Procedure: Blood draw — The following study-specific parameters will be tested: neuropeptide Y 1-36, neuropeptide Y 3-36, total plasma metanephrines, metabolomics analysis
  Time points for blood draw: at admission (routine), 3h (routine), 24h (routine), 48h, 72h and 3 months.
Procedure: Urine (collection over 24h) — The following study-specific parameters will be tested: catecholamines.
  Time points for collection: at 24h, 72h, and 3 months

SUMMARY:
Acute ischemic stroke is caused by blockage of blood vessels in the brain. Blood vessels can be obstructed by several different mechanisms and identification of this cause is essential to minimize the risk of recurrence.

DETAILED DESCRIPTION:
Acute ischemic stroke is caused by blockage of blood vessels in the brain. This obstruction may be due to the presence of a blood clot, which prevents the passage of blood. Because the brain is under-irrigated, nerve cells lack oxygen and nutrients and can die, which can lead to brain function disorder.

Blood vessels can be obstructed by several different mechanisms and identification of this cause is essential to minimize the risk of recurrence. For instance, it may be a blood clot that originally formed in the heart, which breaks off and is carried away by the blood flow into an artery of the brain, which it blocks. The formation of such a clot can be caused by a heart attack, as a heart attack causes reduced mobility of certain parts of the heart, which greatly increases the risk of clot formation. At the same time, a stroke can also induce cardiac changes, for example because of the production of stress hormones secreted during a stroke. These cardiac changes due to stress hormones can greatly look like cardiac changes caused by a heart attack.

As a consequence, when a stroke is caused by a heart attack, it is often very difficult to correctly diagnose the heart attack and therefore treat patients properly. Indeed, symptoms and effects of a stroke and a heart attack may be similar, although these are two completely different medical problems. In order to gain additional knowledge, the investigators aim with this study to make the diagnosis of a heart attack more precise in patients suffering from a stroke.

Hypothesis, primary and secondary objectives:

The investigators postulate that the combination of laboratory, clinical, radiological, echocardiographic and electrophysiological assessments in a predictive score can distinguish myocardial infarction (MI) and neurogenic stunned myocardium (NSM) in stroke patients (MI and NSM defined by cardiac MRI and coronary angiography).

Primary objectives: The primary objective is to assess the prevalence of MI and NSM, with or without wall motion abnormalities, in stroke patients.

Secondary objectives: Secondary objectives aim to develop a predictive score out of laboratory, clinical, radiological (brain MRI), echocardiographic and electrophysiological parameters to identify stroke patients with MI and to distinguish them from patients with NSM.

The project will add important information to the pathogenesis of NSM, the importance of MI in stroke and the clinically relevant question of the management of stroke patients with hsTnT elevations. On one hand, the project offers the chance to improve the identification of patients with relevant coronary sclerosis. The investigators postulate that most of these patients are not identified by current practice. An early identification of these patients is necessary for early treatment and prevention of cardiac events.

On the other hand, the project offers the chance to improve the identification of patients with NSM and to deliver information on clinical relevance of NSM including arrhythmias and wall motion abnormalities. Given the negative association of NSM with outcome after stroke, the identification of NSM patients is the necessary condition for a treatment trial. Beta-blockers could for instance be beneficial for stroke patients with NSM and such a project could have far-reaching consequences on the management of many acute stroke patients in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature.
* Age: ≥ 18 and < 86 years.
* Acute ischemic stroke with symptom onset within 12 hours before admission to hospital.
* Diagnosis of acute ischemic stroke with MRI with diffusion restriction as seen on diffusion weighted imaging.

Exclusion Criteria:

* Pregnancy. A negative pregnancy test upon admission is required for all women with child-bearing potential.
* Standard contraindication for performing MRI.
* Severe renal failure (GFR <40).

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of acute ischemic stroke (< 12 h after symptom onset) confirmed by diffusion weighted MRI will be screened for further inclusion and exclusion criteria.
  This study includes exclusively vulnerable patients, with patients having a life-threatening acute ischemic stroke. The underlying disease needs emergency treatment including immediate management decisions under time pressure. There is no alternative group of patients in whom this study could be performed.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of neurogenic stunned myocardium (NSM) in ischemic stroke patients with elevated hsTnT (≥ 0.015 mg/L) | 48 hours
Prevalence of neurogenic stunned myocardium (NSM) in ischemic stroke patients with elevated hsTnT (≥ 0.015 mg/L) | 3 months

SECONDARY OUTCOMES:
Prevalence of sub(acute) and chronic myocardial infarction in stroke patients with and without elevated hsTnT (≥ 0.015 mg/L) | At baseline, 24 hours, 48 hours, 3 months
Positive and negative predictive value of the developed predictive score to detect myocardial infarction and neurogenic stunned myocardium compared to CMR and coronary angiography | At baseline, 24 hours, 48 hours, 72 hours, 3 months
Influence of neurogenic stunned myocardium on neurological outcome (as measured by modified Rankin Scale) | At baseline, 24 hours, 3 months
  The modified Rankin Scale (mRS) measures the degree of disability or dependence (minimum: 0 [normal]; maximum: 6 [death]). Favorable outcome is defined as a mRS score of 0 to 4, poor outcome as a mRS score of 5 or 6.
Influence of neurogenic stunned myocardium on brain infarct size (as measured by brain MRI) | At baseline, 24 hours, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Simon Jung, PD Dr. med., Study Director — Dep. of Neurology, Inselspital Bern
Locations (1):
- Bern University Hospital - Inselspital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No